

## Consent for participation in research study, neck-specific exercise after whiplash injury

Neck-specific exercise after whiplash injury with problems persisting more than six months. A comparative study of two different forms of exercise: internet-based care combined with a few consultations with a physiotherapist, and a longer period of time exercising at a physiotherapy clinic.

Participation in the study is completely VOLUNTARY, which means that if you choose not to be part of the study this will NOT AFFECT YOUR FUTURE CARE in any negative manner whatsoever. You can terminate your participation at any time.

This document pertains to supplementary investigations with MRI, ultrasound, blood and saliva samples, checks of neck movement and balance tests.

## Participating in the study means that you:

- **Fill out a questionnaire** to ensure that there is nothing to prevent you having an MRI scan.
- Submit blood and saliva samples that are stored in the PAINOMICS biobank.
- **Consent to data being archived** at Linköping University in accordance with applicable archival rules for research data.
- Consent to data collected from the MRI scan being archived in the Region Östergötland image archive. Prior to the imaging material being entered into a computer and analysed, all data is decoded so that no connection to a person can be made. The code key is kept under lock and key and can only be accessed via the project coordinator and project manager. The compilation and reporting of data is carried out in a manner that prevents any connection to any individual being made. All treatment personnel and evaluators are bound by professional confidentiality. The research material is considered to be medical records and is covered by the Secrecy Act.
- Consent to personal data being processed. The data controller is Linköping University via project manager Anneli Peolsson. The data that is processed in the research study is that which is included in the form you fill out prior to the investigation and from the actual MRI scan. You have the right to apply for information and to have any erroneous personal data corrected.
- You can terminate your participation in the study at any point.

Your responses and your results will be processed in a way that prevents any unauthorised persons from accessing them and are covered by the Secrecy Act. There is an insurance policy with the Legal, Financial and Administrative Services Agency via Linköping University. Compensation is paid for long-distance travel (taxable in accordance with the regulations) but not for loss of income.



The project manager for the study is licensed physiotherapist Professor Anneli Peolsson, Department of Medical and Health Sciences (IMH), Division of Physiotherapy, Linköping University.

If you have any questions regarding the MRI scan please contact biomedical engineer and PhD student Anette Karlsson, anette.k.karlsson@liu.se, radiographer Johan Kihlberg, PhD, johan.kihlberg@cmiv.liu.se

If you have questions regarding the questionnaire, ultrasound registration or blood or saliva samples, please contact licensed physiotherapist Gunnel Peterson, PhD, gunnel.peterson@liu.se.

## The research study is carried out with Linköping University as the accountable authority

The research subject has been informed, given the opportunity to ask questions, had them answered and consented to participate in the study as well as to personal data being processed and samples being saved in a biobank.

I have received and understood both oral and written information.

I want to participate in:

- Study regarding MRI scan of the neck Study regarding MRI scan of the brain
- Study regarding ultrasound registration of neck muscles
- Study regarding the neck's movement/proprioception
- Study regarding balance

I understand that participation is voluntary and that I have the right to terminate my participation if I wish to do so.

| Place and date: |
|-----------------------------|
| Personal identity number: |
| Signature: |
| Clarification of signature: |





| Name of researcher that has inform | med me about the |
|------------------------------------|------------------|
| study | |

If you want to withdraw your consent please contact Gunnel Peterson, <a href="mailto:gunnel.peterson@liu.se">gunnel.peterson@liu.se</a>.

The participant keeps the information and receives a copy of the consent form.